CLINICAL TRIAL: NCT04145999
Title: Association of Photobiomodulation With Platelet Rich Plasma Intradermal Injection for Facial Rejuvenation: Controlled, Randomized Clinical Trial
Brief Title: Association of Photobiomodulation With Platelet Rich Plasma Intradermal Injection for Facial Rejuvenation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Erick
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Wrinkle
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A single researcher will perform the treatment and he/she will not perform any evaluation. Pre- and post-treatment evaluations will be made by four examiners (three plastic surgeons and one pathologist) who will not be aware of the group to which each patient will be allocated. Participants will not be aware of whether or not they have received the PRP, the application syringes will be camouflaged with opaque adhesive on the outside and they will not be aware whether or not they have received the PBM application as they will be using eye protection and the person who applies it will position the equipment at the irradiation sites on all participants and will only turn on the light in the specific experimental group. The characteristic sound of the device will be triggered by recording in the placebo groups for the PBM.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP + PBM group (Experimental): This group will receive both PRP application and photobiomodulation.
  Interventions: Procedure: PRP application; Radiation: Photobiomodulation
- PRP + placebo PBM (Experimental): This group will receive PRP application and placebo photobiomodulation.
  Interventions: Procedure: PRP application; Other: Placebo Photobiomodulation
- PBM + placebo PRP (Experimental): This group will receive placebo PRP application with a saline solution and active photobiomodulation.
  Interventions: Other: Placebo PRP application; Radiation: Photobiomodulation

INTERVENTIONS:
Procedure: PRP application — The study participant will receive topical anesthesia with lidocaine ointment (50mg/g). After 5 minutes the face will be cleaned with 0.5% alcohol chlorhexidine solution. The newly obtained platelet-rich plasma activated with 10% calcium chloride packed in a 5mL syringe will be applied to the face using a 30G needle in the frontal, lateral periorbital, nasogenian sulcus, bilateral malar region and an infra-auricular point. 0.1ml per cm2 will be injected, totaling 43 points. Only one application of PRP will be performed at the defined points.
  Arms: PRP + PBM group; PRP + placebo PBM
Other: Placebo PRP application — Blood collection will be performed normally, the time between collection and application of saline will be the same as the PRP protocol, but in this case, the blood will be discarded, only a sample to quantify the number of platelets will be sent for analysis.
  Arms: PBM + placebo PRP
Radiation: Photobiomodulation — Photobiomodulation will be applied with a Cosmedical LED face mask (São Paulo, Brazil) containing 92 red LEDs. The applications will occur in the experimental periods of 0, 3, 7, 14, 21 and 28 days after the application of PRP or placebo.
  Arms: PBM + placebo PRP; PRP + PBM group
Other: Placebo Photobiomodulation — Participants will not be aware of whether or not they have received the PBM application as they will be using eye protection and the researcher will position the equipment at the irradiation locations on all participants. The characteristic sound of the device will be triggered by recording in the placebos groups for the PBM. The placebo applications will occur in the experimental periods of 0, 3, 7, 14, 21 and 28 days after the application of PRP.
  Arms: PRP + placebo PBM

SUMMARY:
Skin aging is an irreversible, slow and progressive process. It is influenced mainly by age, but also by external factors such as ultraviolet radiation, smoking, alcohol, among others. It is increasingly common to look for procedures that slow this process by limiting or hiding its effects on the skin and its appearance. Intradermal platelet-rich plasma (PRP) injection is a new modality of treatment which has possible beneficial effects on skin rejuvenation. In addition, studies have shown photobiomodulation (PBM) benefits to the skin. The purpose of this paper is to investigate the effects of combined use of intradermal PRP injection on the face and photobiomodulation for facial rejuvenation. To this end, a randomized, double-blind, controlled clinical trial will be conducted with volunteer participants who wish to improve facial aesthetics, attended at the Nove de Julho University specialty medical outpatient clinic in the city of São Paulo. Participants will be divided into three groups: one group will undergo intradermal application of PRP in association with PBM; another group will undergo intradermal application of PRP and placebo light and a third group will receive intradermal application of 0.9% saline solution (placebo) associated with PBM. Only one application of PRP or saline solution will be performed at defined points on the face. PBM sessions will be held immediately after the first application of PRP or saline solution, 3 days after the first application and weekly for the next 3 weeks. The following variables will be studied for further analysis: face moldings analyzed by optical coherence tomography; skin viscoelasticity; histological study of the dermis; evolutionary comparison of photographic images by plastic surgeons (Wrinkle Assessment Scale) and participants' satisfaction level (FACE-Q). All data will be statistically evaluated according to their distribution.

ELIGIBILITY:
Inclusion Criteria:

* Menopause (at least 12 months without menstruation);
* Healthy;
* Skin phototype from I to IV by Fitzpatrick classification.

Exclusion Criteria:

* History of photosensitivity;
* Use of corticosteroids, anticoagulants, or any drug known to increase photosensitivity, including systemic retinoids and topical retinoic acid use for the past 6 months;
* Carriers of any collagen-related diseases, malnutrition, anemia, immunosuppression, cancer diseases, smokers, predisposition to hypertrophic and keloid scarring, history of dermatological diseases, facial surgery, facial trauma, conditions that could affect skin condition and psychiatric diseases;
* Patients with blood dyscrasias and thrombocytopenia;
* Esthetic procedures on the face, such as botulinum toxin application in the last year, facial filling in the last 2 years, chemical peels, ablative laser and dermabrasion in the last year;
* Those who do not comply with post-treatment recommendations or fail to attend a treatment session;
* During the procedures those who present any type of complication (hematoma, allergies) will not be part of the statistical analysis, as these cases will not be in the expected pattern for these procedures. However, these data will be described and discussed, as well as possible adverse effects ,and participants will receive treatment to solve the condition.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2020-12-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in Photographic Analysis | Baseline, 3 months and 6 months after treatment.
  Digital photographs of the face obtained before and after 3 and 6 months will be analyzed by 3 plastic surgeons. Each evaluator will receive the same image of wrinkles, all at the end of the experiment. There will be 15 standardized photographs of the face per patient over 6 months of study, totaling 1440 images for each evaluator. Each image should be scored from 0 to 5 using the Wrinkle Assessment Scale.

SECONDARY OUTCOMES:
Change in Optical Coherence Tomography (OCT) Analysis | Baseline, 3 months and 6 months after treatment.
  Negative silicone molds of frontal wrinkles, bilateral periorbital wrinkles and nasolabial folds will be analyzed before treatment and after 3 and 6 months. The parameters to be analyzed are: average surface roughness; average roughness and maximum profile height.
Change in Skin Viscoelasticity | Baseline and 3 months after treatment.
  It will be evaluated in the periocular and bilateral malar region by CUTOMETER DUAL MPA 580® (CK ELETRONIC). The ability of the skin to return to its original position is translated into a measure of elasticity using the device's own software.
Change in Histological Analysis | Baseline and 6 months after treatment.
  Analysis that will be performed by the same pathologist before and after 6 months of treatment. The following parameters will be quantified and compared: epidermal dermal junction length; number of fibroblasts per papillary dermis area; number of blood vessels per basement membrane area; density of collagen fibers by area and density of elastic fibers by area.
Change of Satisfaction with Facial Appearance | Baseline, 3 months and 6 months after treatment.
  Participants will answer the FACE-Q questionnaire, that ranks Satisfaction with Facial Appearance.